CLINICAL TRIAL: NCT06155643
Title: EKO SENSORA: Detecting Clinically Significant Murmurs
Acronym: EkoNM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1635
Record Dates: First submitted 2023-10-31; First posted 2023-12-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Heart Murmurs
Keywords: eko; heart murmur; ai; machine learning; heart murmur detection
MeSH Terms: conditions — Heart Murmurs

STUDY DESIGN:
Intervention Model Description: Use of the Eko device
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Eko Device (Other): Patients with cardiac risk factors
  Interventions: Device: Eko Sensora

INTERVENTIONS:
Device: Eko Sensora — The exam involves placing the stethoscope in the aortic, pulmonic, tricuspid, and mitral areas for 15-30 seconds until a green light is displayed indicating that useful sound has been recorded. The recording is then uploaded by the device using wi-fi to the AI program for analysis. It does not carry patient identifiers. The device then indicates whether a clinically significant heart murmur was heard, and if so in which recording.

SUMMARY:
The Eko Artificial Intelligence (AI) has primarily been evaluated in the primary care setting. The digital stethoscope records a phonocardiogram of heart sounds of the patient and uses machine learning artificial intelligence to identify if there are abnormalities present (Eko Health, 2023).

The Eko SENSORA will be tested in the emergency department. Chest pain, fatigue, shortness of breath and syncope are all symptoms that could indicate a cardiac dysfunction.

The hypothesis is that this device will allow us increased ability to detect valvular heart disease that is clinically significant.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of chest pain, shortness of breath, difficulty breathing, or syncope/near-syncope.
* Patients with chief complaint of Weakness would be eligible if over the age of 50 and have a history of at least two of hypertension, BMI>/= 30, diabetes, hyperlipidemia, atrial fibrillation, heart attack, stroke/Transient ischemic attack, prior cardiac surgery or angiography

Exclusion Criteria:

* Contact isolation patients
* Pediatric patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-07-26 (Estimated)

PRIMARY OUTCOMES:
Number of new clinically significant heart murmurs detected | through study completion, an average of 90 days

SECONDARY OUTCOMES:
Number of echocardiograms ordered | through study completion, an average of 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Corewell Health Lakeland, Saint Joseph, Michigan, United States